CLINICAL TRIAL: NCT02664259
Title: Ultrathin Bronchoscopy With Virtual Bronchoscopic Navigation and Endobronchial Ultrasound for the Diagnosis of Peripheral Pulmonary Lesions Without Fluoroscopy: a Randomized Controlled Trial
Brief Title: UTB-VBN-EBUS With or Without Fluoroscopy for the Diagnosis of PPLs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Jiayuan Sun, Director, Department of Endoscopy, Shanghai Chest Hospital, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SHCHE201602
Record Dates: First submitted 2016-01-22; First posted 2016-01-27 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Lung Cancer
Keywords: Endobronchial ultrasonography; Peripheral pulmonary lesions; Ultrathin bronchoscopy
MeSH Terms: conditions — Lung Neoplasms | interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- UTB-VBN-EBUS group (Experimental): Bronchoscopes with a 3.0-mm distal end diameter and a 1.7-mm working channel diameter are used (BF-Y0058;Olympus).The EBUS probe is confirmed to reach the lesion by EBUS images alone, cytologic and pathologic specimens are obtained without fluoroscopic guidance.
  Interventions: Procedure: VBN; Procedure: EBUS
- UTB-VBN-EBUS-X-ray group (Active Comparator): Bronchoscopes with a 3.0-mm distal end diameter and a 1.7-mm working channel diameter are used (BF-Y0058;Olympus).The EBUS probe is confirmed to reach the lesion by EBUS images and radiograph fluoroscopy, cytologic and pathologic specimens are obtained under fluoroscopic guidance.
  Interventions: Procedure: VBN; Procedure: EBUS; Procedure: X-ray

INTERVENTIONS:
Procedure: VBN — VBN is carried out by a VBN software（DirectPath;Olympus,Japan) which can automatically create virtual bronchoscopic images.
Procedure: EBUS — EBUS is performed using an endoscope ultrasound system , which is equipped with a 20-MHz mechanical radial-type probe (UM-S20-17S;Olympus) with an external diameter of 1.4 mm.
Procedure: X-ray — The radiograph fluoroscopy is performed when the probe is confirmed to reach the lesion by EBUS image ,cytologic and pathologic specimens are obtained under fluoroscopic guidance.
  Arms: UTB-VBN-EBUS-X-ray group

SUMMARY:
The purpose of this study is to evaluate the feasibility,efficacy and safety of ultrathin bronchoscopy(UTB) combined with virtual bronchoscopic navigation(VBN) and endobronchial ultrasound(EBUS) for the diagnosis of peripheral pulmonary lesions (PPLs) without radiographic fluoroscopy.

DETAILED DESCRIPTION:
The investigators evaluate feasibility,efficacy and safety of UTB combined with VBN and EBUS for the diagnosis of PPLs without radiographic fluoroscopy.Bronchoscopes with a 3.0-mm distal end diameter and a 1.7-mm working channel diameter are used (BF-Y0058;Olympus).The final diagnoses are established by pathological evidence from biopsy or cytology specimen including bronchoscopy or other procedures,microbiological analysis and clinical follow-up.The study is designed as a single center prospective randomized controlled trial.The participating center is Department of endoscopy, Shanghai Chest Hospital, Shanghai Jiao Tong University, China.Subjects will be randomized (1:1) to UTB-VBN-EBUS-X-ray group and UTB-VBN-EBUS group based on a randomization schedule.The study is expected to enroll 200 patients with 100 patients of each group.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with peripheral pulmonary lesions suspected to be cancer that need pathologically confirmed;
2. Presence of bronchus leading to or adjacent to the lesion from CT scan.

Exclusion Criteria:

1. Pure ground glass opacity (GGO) lesions;
2. Refusal of participation;
3. Severe cardiopulmonary dysfunction and other indications that can't receive bronchoscopy;
4. Presence of concomitant endobronchial lesion during the brochoscopy procerdure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
The difference of diagnostic value of UTB-VBN-EBUS with fluoroscopy as compared to UTB-VBN-EBUS alone | Up to half year
  The diagnostic value means diagnostic yields in two groups for benign and malignant lesions

SECONDARY OUTCOMES:
The difference of the operation time of UTB-VBN-EBUS with fluoroscopy as compared to UTB-VBN-EBUS alone | Up to half year
  The operation time means the total operation time and the total EBUS time.

OTHER OUTCOMES:
The difference of complications of UTB-VBN-EBUS with fluoroscopy as compared to UTB-VBN-EBUS alone | Up to half year
  Complications mean a composite of operation-related serious adverse events (pneumothorax,bleeding,etc.) during and after the operation in two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, PhD, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Kurimoto N, Miyazawa T, Okimasa S, Maeda A, Oiwa H, Miyazu Y, Murayama M. Endobronchial ultrasonography using a guide sheath increases the ability to diagnose peripheral pulmonary lesions endoscopically. Chest. 2004 Sep;126(3):959-65. doi: 10.1378/chest.126.3.959. PMID 15364779
- [Background] Yoshikawa M, Sukoh N, Yamazaki K, Kanazawa K, Fukumoto S, Harada M, Kikuchi E, Munakata M, Nishimura M, Isobe H. Diagnostic value of endobronchial ultrasonography with a guide sheath for peripheral pulmonary lesions without X-ray fluoroscopy. Chest. 2007 Jun;131(6):1788-93. doi: 10.1378/chest.06-2506. PMID 17565021
- [Background] Steinfort DP, Khor YH, Manser RL, Irving LB. Radial probe endobronchial ultrasound for the diagnosis of peripheral lung cancer: systematic review and meta-analysis. Eur Respir J. 2011 Apr;37(4):902-10. doi: 10.1183/09031936.00075310. Epub 2010 Aug 6. PMID 20693253
- [Background] Oki M, Saka H, Ando M, Asano F, Kurimoto N, Morita K, Kitagawa C, Kogure Y, Miyazawa T. Ultrathin Bronchoscopy with Multimodal Devices for Peripheral Pulmonary Lesions. A Randomized Trial. Am J Respir Crit Care Med. 2015 Aug 15;192(4):468-76. doi: 10.1164/rccm.201502-0205OC. PMID 26039792
- [Background] Ishida T, Asano F, Yamazaki K, Shinagawa N, Oizumi S, Moriya H, Munakata M, Nishimura M; Virtual Navigation in Japan Trial Group. Virtual bronchoscopic navigation combined with endobronchial ultrasound to diagnose small peripheral pulmonary lesions: a randomised trial. Thorax. 2011 Dec;66(12):1072-7. doi: 10.1136/thx.2010.145490. Epub 2011 Jul 11. PMID 21749984
- [Background] Asano F, Shinagawa N, Ishida T, Shindoh J, Anzai M, Tsuzuku A, Oizumi S, Morita S. Virtual bronchoscopic navigation combined with ultrathin bronchoscopy. A randomized clinical trial. Am J Respir Crit Care Med. 2013 Aug 1;188(3):327-33. doi: 10.1164/rccm.201211-2104OC. PMID 23600452